CLINICAL TRIAL: NCT01734421
Title: Efficacacy of a Mobile Application in the Smoking Cessation Among Young Poeple: Cluster Randomized Trial
Brief Title: Efficacy of a Mobile Application in the Smoking Cessation Among Young People
Acronym: TOBB_STOP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Fundacio d'Investigacio en Atencio Primaria Jordi Gol i Gurina (Other)
Collaborators: Preventive Services and Health Promotion Research Network (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PI12/01977
Record Dates: First submitted 2012-11-22; First posted 2012-11-27 (Estimated); Last update posted 2012-11-27 (Estimated); Status verified 2012-11

CONDITIONS: Smoking Cessation
Keywords: Smoking cessation; Primary health care; Young people; Cellular phone
MeSH Terms: conditions — Smoking Cessation | interventions — Control Groups

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (2):
- Control group (Other): Habitual deshabituation in the control group following the guidelines of the primary health care institution.
  Interventions: Other: Control group
- Cell phone Aplication for Smarth Phone (Active Comparator): Cell phone 6-month implementation of recommendations of a Clinical Practice Guideline smoking cessation which includes mobile APPs application
  Interventions: Device: Cell phone Aplication for Smarth Phone

INTERVENTIONS:
Other: Control group — 6-month implementation of recommendations of a Clinical Practice Guideline smoking cessation
  Arms: Control group
Device: Cell phone Aplication for Smarth Phone
  Arms: Cell phone Aplication for Smarth Phone

SUMMARY:
AIM: To assess the efficacy of an intervention based on the specific design and implementation of a mobile application (APP) in order to reduce the prevalence of smoking consumption among young people motivated 18 to 30 years METHODS: Cluster randomised clinical trial. Unit of randomization: Primary Health Care Centers (PHCC). Intention to treat analysis. STUDY POPULATION: Motivated young smokers of 10 or more cigarettes per day aged 18 to 30 years consulting for any reason to PHCC and who provided written informed consent to participate in the trial.

INTERVENTION: 6-month implementation of recommendations of a Clinical Practice Guideline smoking cessation which includes mobile APPs application. Control group: usual care. OUTCOME MEASURES: Abstinence at 12 months confirmed by exhaled air carbon monoxide concentration of less or iqual 10 parts per million in each control.

RESULTS: The application of a smoking cessation intervention with a mobile APPs application will improve the smoking cessation success rate in smokers, besides of their intention or not to give up smoking at baseline.

ELIGIBILITY:
Inclusion Criteria:

* Participant between 18 t0 30 years old smoking 10 or more cigarretes at day
* To have a smarthphone (Android, ios Ihpone, ios Ipad)
* Normal and high motivation for smocking cessation

Exclusion Criteria:

* To have other addictions
* Participants with Blackberry smarthphone

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 604 (Estimated)
Dates: Start 2013-01; Primary Completion 2015-06 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Smoking cessation | Change in smoking status from baseline at 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Jordi Gol i Gurina Foundation, Barcelona, Spain

REFERENCES:
- [Derived] Palleja-Millan M, Rey-Renones C, Barrera Uriarte ML, Granado-Font E, Basora J, Flores-Mateo G, Duch J. Evaluation of the Tobbstop Mobile App for Smoking Cessation: Cluster Randomized Controlled Clinical Trial. JMIR Mhealth Uhealth. 2020 Jun 26;8(6):e15951. doi: 10.2196/15951. PMID 32589153
- [Derived] Marin-Gomez FX, Garcia-Moreno Marchan R, Mayos-Fernandez A, Flores-Mateo G, Granado-Font E, Barrera Uriarte ML, Duch J, Rey-Renones C. Exploring Efficacy of a Serious Game (Tobbstop) for Smoking Cessation During Pregnancy: Randomized Controlled Trial. JMIR Serious Games. 2019 Mar 27;7(1):e12835. doi: 10.2196/12835. PMID 30916655
- [Derived] Valdivieso-Lopez E, Flores-Mateo G, Molina-Gomez JD, Rey-Renones C, Barrera Uriarte ML, Duch J, Valverde A. Efficacy of a mobile application for smoking cessation in young people: study protocol for a clustered, randomized trial. BMC Public Health. 2013 Aug 1;13:704. doi: 10.1186/1471-2458-13-704. PMID 23915067